CLINICAL TRIAL: NCT06341140
Title: Does Individualized Breastfeeding Support Make a Difference in Exclusive Breastfeeding, Breast Problem Occurrence, and Breastfeeding Self-Efficacy in the First 6 Months: Randomized Controlled Study
Brief Title: The Effect of Breastfeeding Support on Exclusive Breastfeeding, Occurrence of Breast Problems and Breastfeeding Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Collaborators: Manisa Celal Bayar University (Other)
Responsible Party: Principal Investigator, Seçil Köken Durgun, Principal Investigator, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: secil koken
Record Dates: First submitted 2024-02-29; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Experimental): Pregnant women in the control group were given a booklet containing information about breastfeeding. In the postpartum period, the breastfeeding process was observed with home visits and telephone for the first 6 months.
  Interventions: Other: Booklet containing information about breastfeeding
- intervention (Experimental): Pregnant women in the intervention group were given a booklet containing information about breastfeeding. At the same time, individual breastfeeding support was provided with a wearable breastfeeding model. In the postpartum period, the breastfeeding process was observed with home visits and telephone for the first 6 months.
  Interventions: Other: Breastfeeding support and Booklet containing information about breastfeeding

INTERVENTIONS:
Other: Breastfeeding support and Booklet containing information about breastfeeding — Pregnant women in the intervention group were given individual counseling with a wearable breastfeeding model. During postnatal home visits, mothers were given support on breastfeeding, breast problems were addressed, and information was given to support the mother's self-efficacy.
  Arms: intervention
Other: Booklet containing information about breastfeeding — Pregnant women in the control group were given only a breastfeeding booklet, breastfeeding status, breast problems and breastfeeding self-efficacy were evaluated during postnatal home visits and telephone interviews, and risky situations were referred to health professionals.
  Arms: control

SUMMARY:
The aim of the study is to determine the effect of individual breastfeeding support on the lactation process. The research is a randomized controlled experimental study. The sample of the study consisted of pregnant women who applied to the Obstetrics Polyclinic of a university hospital (intervention=51, control=51). In the study, individual breastfeeding education was given to the intervention group during the antenatal period, and a training booklet was given to the control group. In the postpartum period, home visits and phone follow-ups were carried out for both groups between the fifth day and the sixth month. The effect of breastfeeding counseling on the lactation process; The duration of exclusive breastfeeding, breast problems and breastfeeding success was evaluated with. The data of the study were collected using the Pregnant, Postpartum-Newborn Information Form, Breastfeeding Questionnaire, Breast Problems Diagnosis Form, LATCH Breastfeeding Diagnostic Tool and Breastfeeding Self-Efficacy Scale.

ELIGIBILITY:
İnclusion Criteria:

* Open communication and collaboration
* Over 18 years of age
* Having a singleton pregnancy
* Never given birth,
* At least in the 35th week of gestation,
* Residing in Manisa Central districts (Yunusemre and Şehzadeler),
* There is no maternal obstacle that would affect breastfeeding,
* Having no vision or hearing problems,
* Those who are willing to participate in the study

Exclusion Criteria:

* At the beginning of the research;
* Under 18 years of age,
* Having a risky pregnancy,
* Having breastfeeding experience,
* Less than the 35th gestational week,
* Residing outside Manisa Central districts (Yunusemre and Şehzadeler),
* Any maternal disability that may affect breastfeeding,
* Pregnant women who did not want to participate in the study were excluded.

During the research process;

* Those who want to leave the job,
* If the baby has any obstacle that may affect breastfeeding (presence of anomaly, stay in intensive care, etc.),
* Cannot be reached within the first 5 days after birth,
* Mothers who changed their residence to live in another city/district other than Manisa Central districts (Yunusemre and Şehzadeler) were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Situation of mothers feeding their babies exclusively with breast milk | 6 months
  Determination of mothers' status of exclusively breastfeeding their babies for the first 6 months using a survey form created by researchers.
Mothers experiencing breast problems | 6 months
  Determination of breast problems that occur during the breastfeeding process with a survey created by researchers.
Determination of mothers' breastfeeding self-efficacy | 6 months
  Breastfeeding competencies were assessed with the LATCH breastfeeding diagnostic tool and the breastfeeding self-efficacy scale. Mothers' breastfeeding success was examined with the LATCH breastfeeding diagnostic tool. On this scale, they can get a minimum of 0 and a maximum of 10 points. As the score increases, breastfeeding success increases. The breastfeeding self-efficacy scale determines the self-efficacy of mothers and can get a minimum of 33 and a maximum of 165 points. As the average score increases, breastfeeding self-efficacy is expressed as high.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Cambaz Ulaş, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)